CLINICAL TRIAL: NCT02310841
Title: Pilotstudie zu Patientenkooperativen Regelungsstrategien für Aktuierte Oberschenkelexoprothesen
Brief Title: Pilot Study for Patient-cooperative Control Strategies for Actuated Transfemoral Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Verena Klamroth, MD, Swiss Federal Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KEK-ZH-2013-0034; 2013-MD-0004 (Other: Swissmedic)
Record Dates: First submitted 2014-10-29; First posted 2014-12-08 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-12

CONDITIONS: Gait Disorder, Sensorimotor
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- unilateral transfemoral amputees (Experimental)
  Interventions: Device: ANGELAA

INTERVENTIONS:
Device: ANGELAA — Different control strategies with transfemoral prosthesis prototype ANGELAA, developed at the Sensory-Motor Systems Lab, ETH Zurich, not commercially available, only 1 device exists

SUMMARY:
This pilot study investigates the feasibility of novel control strategies for actuated transfemoral prostheses. Several parameters from gait analysis (including motion-capture and ground reaction force measurements) are analyzed. The subjective perception of prosthetic functionality is captured with a questionnaire.

DETAILED DESCRIPTION:
Setting of the study: Conventional prostheses for transfemoral amputees are mostly simple mechanic joints, or have micro-processor-controlled damping. The prototype tested in this study is equipped with a motor that can actively move the knee joint. Therefore, movements like, for example, alternating stair climbing, are possible that cannot be realized with pure mechanical and actively damped prostheses. During level-ground walking, it is hypothesized that less compensatory movements are needed. We have developed an actuated prototypical prosthesis and new control strategies which should facilitate both level-ground walking and stair climbing. Parts of the control strategies have been tested in able-bodied subjects [1]. This control strategy has been extended such that only biological stiffness modulation can be rendered [2].

Hypothesis: Subjects can use our transfemoral prosthesis to walk on level-ground, to climb several steps and to overcome small obstacles without prior training. The user-cooperative control is intuitive and easily learnable.

Objective of the study: This pilot study is meant to investigate the general feasibility of novel control strategies for actuated transfemoral prostheses. Parameters of a standard gait analysis, like ground reaction forces and kinematics (using a motion capture system), will be recorded. From this data, gait symmetry, step length, walking speed, and other measures can be calculated. The subjective impression of the user will be evaluated with a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Written consent of participant
* For amputees: regular use of a transfemoral prosthesis
* For amputees: transfemoral amputation

Exclusion Criteria:

* Bodymass > 100 kg
* For amputees: mobility class 1
* For amputees: no stable residual leg volume
* For amputees: constrictive contractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change of gait pattern using an actuated transfemoral prosthesis compared to a passive prosthesis | Subjects will come to the gait lab for two days. The experiment itself lasts about 1.5 hours per day.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, Prof. Dr, Principal Investigator — Sensory Motor Systems Lab, ETH Zurich
Locations (1):
- University Hospital Balgrist, Zurich, Switzerland